CLINICAL TRIAL: NCT06106750
Title: The Efficacy and Safety of Endoscopic Scissors Cutting Nasobiliary Ducts in the Treatment of Malignant Hilar Biliary Tract Stenosis
Brief Title: Endoscopic Scissors Cutting Nasobiliary Duct VS Bilateral Plastic Stent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Department director, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-10
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Cholangiocarcinoma, Hilar; Biliary Stricture; Hilar Cholangiocarcinoma; Klatskin Tumor; Biliary Disease; Bile Duct Diseases; Bile Duct Stenosis
Keywords: Endoscopic Retrograde Cholangiopancreatography; Nasobiliary Duct; Stent; Endoscopic Drainage
MeSH Terms: conditions — Klatskin Tumor; Gallbladder Diseases; Bile Duct Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasobiliary duct cutting (Experimental): Endoscopic retrograde cholangiopancreatography and endoscopic nasobiliary duct placement and drainage are conducted first. Upon achieving a postoperative state marked by satisfactory nasobiliary duct drainage and overall patient stability, the procedure entails the employment of endoscopic scissors. The tools are applied to make an incision on the external segment of the nasobiliary duct, positioned beyond the aperture of the primary duodenal papilla. Then, extracting the severed nasobiliary duct and retaining the portion inside it.
  Interventions: Device: Endoscopic nasobiliary duct cutting
- Bilateral plastic stent (Active Comparator): Standard protocol for the placement of bilateral biliary plastic stents in the management of malignant hilar biliary tract stenosis
  Interventions: Device: Bilateral plastic stent

INTERVENTIONS:
Device: Endoscopic nasobiliary duct cutting — Endoscopic retrograde cholangiopancreatography and endoscopic nasobiliary duct placement and drainage are conducted first. Upon achieving a postoperative state marked by satisfactory nasobiliary duct drainage and overall patient stability, the procedure entails the employment of endoscopic scissors. The tools are applied to make an incision on the external segment of the nasobiliary duct, positioned beyond the aperture of the primary duodenal papilla. Then extracting the severed nasobiliary duct and retaining the portion inside the duct.
  Arms: Nasobiliary duct cutting
Device: Bilateral plastic stent — Standard protocol for the placement of bilateral biliary plastic stents in the management of malignant hilar biliary tract stenosis
  Arms: Bilateral plastic stent

SUMMARY:
The purpose of this study is to explore the efficacy and safety of endoscopic scissors cutting nasobiliary ducts in the treatment of malignant hilar biliary tract stenosis

DETAILED DESCRIPTION:
The early diagnosis of hilar bile duct stenosis is difficult, and when the patient is diagnosed, the opportunity for surgical radical resection is lost, resulting in a poor prognosis. Effective palliative treatment can significantly improve their quality of life and survival time. The method of cutting nasobiliary ducts with endoscopic scissors has many advantages. Firstly, there are multiple lateral foramen of the nasobiliary duct, which increases the drainage area. Secondly, the nasobiliary duct can be retained in the secondary bile duct, which is difficult to achieve with a conventional stent. The use of nasobiliary ducts can also reduce the difficulty of converting from external drainage to internal drainage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old and under 80 years old who were planned to carry out ERCP for malignant hilar biliary duct stenosis
2. Clinically and pathologically confirmed malignant hilar biliary duct stenosis
3. MRCP determines Bismuth classification: II-IV type
4. Comply with research procedures and sign the informed consent form

Exclusion Criteria:

1. The patient has multiple organ dysfunction and cannot tolerate endoscopic treatment
2. The patient has undergone biliary drainage (endoscopic, percutaneous, or surgical)
3. The patient is currently suffering from cholangitis
4. The patient is participating in other clinical trials
5. Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of cholangitis | 1 month
  Cholangitis that occurred within 1 month after endoscopic retrograde cholangiopancreatography(ERCP).
Clinical success | 1 month
  Clinical success was defined that the decrease in the total bilirubin level to less than 50% of the pretreatment value within 1 week or to less than 75% within 1 month.

SECONDARY OUTCOMES:
Re-intervention | 6 month
  Re-intervention was defined that endoscopic or percutaneous procedure to improve biliary drainage for jaundice or cholangitis after successful placement.
Adverse events | 1 month
  ERCP-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Yang, Doctor, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kawashima H, Itoh A, Ohno E, Itoh Y, Ebata T, Nagino M, Goto H, Hirooka Y. Preoperative endoscopic nasobiliary drainage in 164 consecutive patients with suspected perihilar cholangiocarcinoma: a retrospective study of efficacy and risk factors related to complications. Ann Surg. 2013 Jan;257(1):121-7. doi: 10.1097/SLA.0b013e318262b2e9. PMID 22895398
- [Result] Kawakami H, Kuwatani M, Onodera M, Haba S, Eto K, Ehira N, Yamato H, Kudo T, Tanaka E, Hirano S, Kondo S, Asaka M. Endoscopic nasobiliary drainage is the most suitable preoperative biliary drainage method in the management of patients with hilar cholangiocarcinoma. J Gastroenterol. 2011 Feb;46(2):242-8. doi: 10.1007/s00535-010-0298-1. Epub 2010 Aug 11. PMID 20700608
- [Result] Hakuta R, Kogure H, Nakai Y, Kawakami H, Maguchi H, Mukai T, Iwashita T, Saito T, Togawa O, Matsubara S, Hayashi T, Maetani I, Ito Y, Hasebe O, Itoi T, Hanada K, Isayama H. Unilateral versus Bilateral Endoscopic Nasobiliary Drainage and Subsequent Metal Stent Placement for Unresectable Malignant Hilar Obstruction: A Multicenter Randomized Controlled Trial. J Clin Med. 2021 Jan 8;10(2):206. doi: 10.3390/jcm10020206. PMID 33430020
- [Result] Sugiura R, Kuwatani M, Hayashi T, Yoshida M, Ihara H, Yamato H, Onodera M, Katanuma A; Hokkaido Interventional EUS/ERCP study (HONEST) group. Endoscopic Nasobiliary Drainage Comparable with Endoscopic Biliary Stenting as a Preoperative Drainage Method for Malignant Hilar Biliary Obstruction: A Multicenter Retrospective Study. Digestion. 2022;103(3):205-216. doi: 10.1159/000521510. Epub 2022 Jan 26. PMID 35081535